CLINICAL TRIAL: NCT01725620
Title: A Randomized, Double-blind, Single-dosing, 2-way Cross-over Study to Compate the Safety and Pharmacokinetic Characteristics of LBEC0101(Etanercept) 25mg With Those of Enbrel® 25mg After Subcutaneous Injection in Healthy Male Volunteers
Brief Title: Study to Compare the Safety and Pharmacokinetic Characteristics of LBEC0101 25mg With Those of Enbrel®
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: LG Life Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: LG-ECCL003
Record Dates: First submitted 2012-11-09; First posted 2012-11-14 (Estimated); Last update posted 2015-01-30 (Estimated); Status verified 2015-01

CONDITIONS: Healthy
MeSH Terms: interventions — LBEC0101; Etanercept

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Group 1 (Experimental): Enbrel, LBEC0101
  Interventions: Drug: LBEC0101 (Etanercept 25mg); Drug: Enbrel (Etanercept 25mg)
- Group 2 (Experimental): LBEC0101, Enbrel
  Interventions: Drug: LBEC0101 (Etanercept 25mg); Drug: Enbrel (Etanercept 25mg)

INTERVENTIONS:
Drug: LBEC0101 (Etanercept 25mg)
Drug: Enbrel (Etanercept 25mg)

SUMMARY:
To compare the pharmacokinetic characteristic of LBEC0101 25mg with active comparator, Enbrel® 25mg.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males, 20 to 45 years of age the moment of screening
* Body mass index is between 18.0 and 30.0 kg/m

Exclusion Criteria:

* The tuberculosis patient of latent tuberculosis patient
* Hypersensitivity response to the test and comparator drugs

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2012-11; Primary Completion 2013-04 (Actual); Study Completion 2014-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kyung-Sang Yu, M.D., Ph.D., Principal Investigator — Seoul National University College of Medicine and Hospitaal
Locations (1):
- Seoul National University Hospital, Clinical Trial Center, Seoul, Seoul, South Korea

REFERENCES:
- [Derived] Lee H, Chung H, Lee S, Lee H, Yang SM, Yoon SH, Cho JY, Jang IJ, Yu KS. LBEC0101, A Proposed Etanercept Biosimilar: Pharmacokinetics, Immunogenicity, and Tolerability Profiles Compared with a Reference Biologic Product in Healthy Male Subjects. BioDrugs. 2017 Aug;31(4):349-355. doi: 10.1007/s40259-017-0230-9. PMID 28551775